CLINICAL TRIAL: NCT01574222
Title: Intratumoral Genetic Therapy for Lung Cancer
Brief Title: A Vaccine Trial for Patients With Stage IIIB, IV, or Recurrent Non-Small Cell Lung Cancer
Acronym: VTNSCLC
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Estimated Primary Completion Date: March 2017 (Final data collection date for primary outcome measure)
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Jonsson Comprehensive Cancer Center (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN-004-09F
Record Dates: First submitted 2012-03-28; First posted 2012-04-10 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Non-Small Cell Lung Cancer (NSCLC)
Keywords: Stages IIIB, IV, and recurrent NSCLC; Carcinoma, Non-small cell lung; Lung Neoplasms; Carcinoma, Bronchogenic; Thoracic Neoplasms; Neoplasms by Site; Neoplasms; Lung Diseases
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Carcinoma, Bronchogenic; Thoracic Neoplasms; Neoplasms by Site; Neoplasms; Lung Diseases

STUDY DESIGN:
Masking Description: No masking
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): Eligible patients will be assigned to a cohort and will receive intratumoral injections of Ad-CCL21-DC in conjunction with tumor sampling
  Interventions: Biological: autologous dendritic cell adenovirus CCL21 vaccine

INTERVENTIONS:
Biological: autologous dendritic cell adenovirus CCL21 vaccine — Eligible patients will be assigned to a cohort and will receive intratumoral injections of Ad-CCL21-DC in conjunction with tumor sampling.
  Other Names: 10-000039, UCLA-NCI 7888, 03-06-008

SUMMARY:
The purpose of this study is to determine the dose that the vaccine can be given safely to patients when injected directly into the lung tumor, without any serious side effects.

DETAILED DESCRIPTION:
Primary

- to determine the safety, toxicity, and Maximum Tolerated Dose (MTD) of autologous dendritic cell-adenovirus chemokine (C-C motif) ligand 21 (CCL21) vaccine administered as an intratumoral injection in treating patients with stage IIIB, IV, or recurrent non-small cell lung cancer

Secondary

* to determine the biologic and clinical responses to therapy
* to determine treatment-related toxicity using the NCI Common Toxicity Criteria
* to identify the maximum tolerated dose (MTD)
* to monitor patients for evidence of autologous dendritic cell-adenovirus CCL21 vaccine-induced cytokines and antigen-specific immune responses
* to detect immune responses to tumor-associated antigens and vector
* to assess patients for objective signs of tumor regression (RECIST criteria)

ELIGIBILITY:
Inclusion Criteria:

Screening, physical exams, blood draws, CT scans, and follow-up will be performed at VA Greater Los Angeles. All interventional procedures including leukapheresis, CT guided/bronchoscopic biopsies and vaccine injections will be performed at University of California Los Angeles (UCLA).

* Adults over the age of 21 capable of giving informed consent
* Pathologically confirmed non-small cell lung cancer (NSCLC)
* Stage IIIB, IV or recurrent disease
* Progressive disease despite one or more prior chemotherapy regimens as standard of care OR patient refusal of standard chemotherapy
* Measurable metastatic disease by RECIST guidelines
* Patients with a major endobronchial lesion in the segmental, lobar, or mainstem bronchus with complete obstruction of the airway may be eligible for bronchoscopic injection provided there is no evidence of respiratory failure (defined as SaO2 at least 90% on room air, PCO2 less than, or equal to 45 mm Hg, or FEV1 greater than 1.0L)
* Patients with an endobronchial lesion in the segmental bronchus with variable stenosis (not completely obstructed) and not amenable to standard palliative airway treatments (i.e., laser and stenting) may be eligible for bronchoscopic injection if there is no indication of respiratory failure as defined above
* Patient with bullous disease may undergo CT-guided transthoracic injection provided the targeted tumor has an intended needle path without crossing bullae
* ECOG performance status 0-2
* BUN less than or equal to 40 OR serum creatinine less than 2 Serum total bilirubin less than or equal to 1.5 OR serum transaminases less than or equal to 2.5 times upper limit of normal (ULN)
* Negative pregnancy test (if applicable)
* Fertile patients must use effective contraception
* More than 14 days since prior acute therapy for viral, bacterial, or fungal infections
* More than 30 days since prior and no concurrent corticosteroids
* More than 15 days since prior radiotherapy
* More than 30 days since prior chemotherapy, or non-cytotoxic investigational agents

Exclusion Criteria:

* Active CNS metastases (i.e., progression of CNS disease during the past 30 days without intervention)
* Evidence of coagulopathy, defined as PT and/or PTT more than 1.5 times ULN or platelets more than or equal to 100,000/mm3.
* Evidence of leukoplakia, defined as absolute neutrophil count more than or equal to 1,500/mm3
* Evidence of respiratory failure (defined as SaO2 less than 90% on room air, PCO2 more than 45 mm Hg, or FEV1 less than 1.0 L
* NYHA class III-IV within the past year
* Myocardial infarction within the past year
* Comorbid disease or medical condition that would impair the ability of the patient to receive or comply with the study protocol
* Acute viral, bacterial or fungal infection that requires specific therapy
* HIV positive
* Hypersensitivity to any reagents used in the study
* Signs or sensitivity of acute adenoviral infection (i.e., conjunctivitis or documented adenoviral upper respiratory infection)
* Pregnant or nursing
* Prior organ allograft

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-10-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 28 Days
  Toxicity as measured by NCI Common Toxicity Criteria

SECONDARY OUTCOMES:
Disease status at days 28 and 56 days | 28 and 56 Days
  Immune response assessment by antigen-specific interferon gamma (IFNy) Enzyme-Linked ImmunoSpot (ELISPOT) assays on days 0, 28, and 56

CONTACTS AND LOCATIONS:
Overall Officials: Steven Dubinett, MD, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee JM, Lee MH, Garon E, Goldman JW, Salehi-Rad R, Baratelli FE, Schaue D, Wang G, Rosen F, Yanagawa J, Walser TC, Lin Y, Park SJ, Adams S, Marincola FM, Tumeh PC, Abtin F, Suh R, Reckamp KL, Lee G, Wallace WD, Lee S, Zeng G, Elashoff DA, Sharma S, Dubinett SM. Phase I Trial of Intratumoral Injection of CCL21 Gene-Modified Dendritic Cells in Lung Cancer Elicits Tumor-Specific Immune Responses and CD8+ T-cell Infiltration. Clin Cancer Res. 2017 Aug 15;23(16):4556-4568. doi: 10.1158/1078-0432.CCR-16-2821. Epub 2017 May 3. PMID 28468947
- See also: Click here for more information about this study: Intratumoral genetic therapy for lung cancer — https://clinicaltrials.gov/ct2/show/NCT00601094